CLINICAL TRIAL: NCT03161483
Title: A PHASE 2, MULTICENTER, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY TO EVALUATE THE EFFICACY AND SAFETY OF CC-220 IN SUBJECTS WITH ACTIVE SYSTEMIC LUPUS ERYTHEMATOSUS
Brief Title: A Study to Evaluate the Efficacy and Safety of CC-220 in Subjects With Active Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-220-SLE-002; U1111-1195-7804 (Registry Identifier: WHO)
Record Dates: First submitted 2017-05-18; First posted 2017-05-19 (Actual); Results first posted 2021-02-18 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: CC-220; Safety; Efficacy; Active Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — iberdomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CC-220 0.45 mg QD Placebo Controlled Phase (Experimental): * At Weeks 0 to 24: CC-220 Placebo Controlled Phase: CC-220 0.45 mg once daily (QD)
  * At Weeks 24 to 52: CC-220 Active Treatment Phase: CC-220 0.45 mg once daily (QD)
  * Long-term Extension Phase (52 weeks to 104 weeks): At Week 52 all subjects who elect to continue in the Long-term Extension will stay on the same dose they were on at the conclusion of the randomized, double-blind, active treatment phase.
  Interventions: Drug: CC-220; Other: Placebo
- C-220 0.3 mg QD Placebo Controlled Phase (Experimental): * At Weeks 0 to 24: CC-220 Placebo Controlled Phase: CC-220 0.3 mg once daily (QD)
  * At Weeks 24 to 52: CC-220 Active Treatment Phase: CC-220 0.30 mg once daily (QD)
  * Long-term Extension Phase (52 weeks to 104 weeks): At Week 52 all subjects who elect to continue in the Long-term Extension will stay on the same dose they were on at the conclusion of the randomized, double-blind, active treatment phase.
  Interventions: Drug: CC-220; Other: Placebo
- CC-220 0.15 mg QD Placebo Controlled Phase (Experimental): * At Weeks 0 to 24: CC-220 Placebo Controlled Phase: CC-220 0.15 mg once daily (QD)
  * At Weeks 24 to 52: CC-220 Active Treatment Phase: CC-220 0.15 mg once daily (QD)
  * Long-term Extension Phase (52 weeks to 104 weeks): At Week 52 all subjects who elect to continue in the Long-term Extension will stay on the same dose they were on at the conclusion of the randomized, double-blind, active treatment phase.
  Interventions: Drug: CC-220; Other: Placebo
- Placebo (Placebo Comparator): Weeks 0 to 24: CC-220 Placebo Controlled Phase: placebo once daily (QD)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CC-220 — CC-220
  Arms: C-220 0.3 mg QD Placebo Controlled Phase; CC-220 0.15 mg QD Placebo Controlled Phase; CC-220 0.45 mg QD Placebo Controlled Phase
Other: Placebo — Placebo QD PO

SUMMARY:
The purpose of this Phase 2, multicenter, randomized, placebo-controlled, double-blind study to evaluate the efficacy and safety of an oral treatment regimen of CC-220 versus placebo in adult subjects with active systemic lupus erythematosus.

Approximately 280 subjects with a documented diagnosis of SLE will be randomized 2:2:1:2 to receive CC-220 (0.45 mg QD, 0.3 mg QD or 0.15 mg QD) or identically appearing placebo.

DETAILED DESCRIPTION:
The study consists of four phases:

* 4-week Screening Phase
* 24-week placebo-controlled phase Subjects will receive either 0.45 mg QD, 0.3 mg QD, 0.15 mg QD or placebo for the first 24 weeks of treatment.
* 28-week active treatment phase At Week 24, all subjects on placebo will be re-randomized to active treatment.
* 52-week long-term extension phase Subjects who complete the treatment phase may be eligible to roll over into a Long-term Extension of up to 52 weeks of treatment.
* 4 - 12-week observational follow-up All subjects who complete 52 weeks of treatment or discontinue the study early will enter a post-treatment observation follow-up phase. The Observational Follow-up Phase will consist of one visit 4 weeks following cessation of study drug for all subjects with an additional 12-week Observational Follow-up visit for males only.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or older at the time of signing the informed consent.
* Have a diagnosis of SLE for at least 6 months prior to the Screening Visit and fulfill the 1997 update of the 1982 American College of Rheumatology (ACR) Classification Criteria for SLE at the Screening Visit.
* A SLEDAI 2K score of ≥ 6 points, WITH at least 4 points being a "clinical" SLEDAI 2K score. The "clinical" score excludes points attributable to any urine or blood laboratory results including immunologic measures.
* At the Baseline Visit, a clinical SLEDAI 2K score of ≥ 4 points.
* Have at least one of the following positive antibodies associated with SLE per the central laboratory within the Screening Phase:

  * Positive antinuclear antibody (ANA) test at the central laboratory with a titer of 1:40 or greater, associated with a diagnosis of SLE,
  * Anti-dsDNA antibodies elevated to above normal
  * Anti-Smith (anti-Sm) antibody elevated to above normal
* Females of childbearing potential must: Have two negative pregnancy tests as verified by the Investigator prior to starting study therapy. She must agree to ongoing pregnancy testing during the course of the study, and after end of study treatment.

  o Either commit to true abstinence from heterosexual contact or agree to use two forms of reliable contraception simultaneously.
* Male subjects must: Practice true abstinence or agree to use a barrier contraception during sexual contact.

All subjects must:

* Understand that the IP could have potential teratogenic risk.
* Agree to abstain from donating blood while taking IP and for 28 days following discontinuation of the IP.

  * Have been treated with at least one of the following SLE medications prior to the Screening Visit: antimalarials, immunosuppressants, and/or corticosteroids.
  * Currently receiving stable doses of at least one of the following medications: systemic corticosteroids, antimalarials, and/or immunosuppressants.

Exclusion Criteria:

* Received intra-articular, intralesional, subcutaneous, intradermal, intramuscular or IV pulse corticosteroids 6 weeks prior to the Baseline Visit.
* Received any other biologic or non-biologic immunosuppressive agent within 2 months of 5 pharmacokinetic half-lives (whichever is longer) prior to the Baseline Visit.
* Have severe lupus nephritis defined as: estimated glomerular filtration rate of < 45 mL/1.73 m2 or proteinuria > 2000 mg/day based on protein to creatinine ratio, or active lupus nephritis that may require 'induction' therapy
* Have active, severe or unstable neuropsychiatric lupus disease within 6 months of the Screening Visit.
* Have serologic tests consistent with infection with either hepatitis B or hepatitis C, and/or confirmed history of hepatitis B or hepatitis C infection.
* Have history of congenital and/or acquired immunodeficiencies (eg, common variable immunodeficiency, human immunodeficiency virus, etc).
* Have active or history of recurrent bacterial, viral, fungal, mycobacterial or other infections, or any major episode of infection requiring hospitalization or treatment with intravenous or oral antibiotics within 4 weeks of the Screening Visit and at any time during the Screening Phase, up through the first dose of IP.
* Have active tuberculosis or a history of latent or active tuberculosis
* Have malignancy or history of malignancy, except for:

  * treated (eg, cured) basal cell or squamous cell in situ skin carcinomas
  * treated (eg, cured) cervical intraepithelial neoplasia Grade 1 and Grade 2
  * treated (eg, cured) carcinoma in situ of the cervix with no evidence of recurrence within 5 years of the Screening Visit.
* Have a diagnosis or history consistent with Antiphospholipid Syndrome or "triple antiphospholipid positivity" (ie, positive lupus anticoagulant, anticardiolipin, and anti-B2 glycoprotein).
* Have history of arterial or venous thrombosis
* Have history or current diagnosis of peripheral neuropathy (sensory or motor) ≥ Grade 2.
* Have presence of active uveitis or any other ophthalmological finding that in the opinion of the Investigator is clinically significant.
* Have other non-SLE driven inflammatory joint or skin disease or overlap syndromes as the primary disease.
* Have clinically significant or unstable or uncontrolled acute or chronic disease not due to SLE
* Does not meet required laboratory criteria.
* Does not meet pre-specified periods for prohibited medications.
* Pregnant or a breast-feeding female.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nataliya Agafonova, MD, Study Director — Celgene Corporation
Locations (184):
- United States (46):
  - Clinical and Translational Research Center of Alabama, PC, Tuscaloosa, Alabama
  - AZ Arthritis and Rheum Rsch, PLLC, Mesa, Arizona
  - Saint Jude Heritage Medical Center, Fullerton, California
  - University of California San Diego Medical Center, La Jolla, California
  - UCLA Division of Rheumatology, Los Angeles, California
  - Desert Medical Advances, Palm Desert, California
  - C Michael Neuwelt M D, San Leandro, California
  - Inland Rheumatology Clinical Trials, Upland, California
  - University of Colorado Denver, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Centre For Rheumatology, Immun. And Arthritis, Fort Lauderdale, Florida
  - University of Florida College of Medicine, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Integral Rheumatology and Immunology Specialists, Plantation, Florida
  - Bay Care Medical Group, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Piedmont Hospital - Atlanta, Atlanta, Georgia
  - Jefrey Lieberman, MD, PC, Decatur, Georgia
  - North Georgia Rheumatology, Lawrenceville, Georgia
  - Clinic of Robert Hozman, Skokie, Illinois
  - University of Maryland - School of Medicine, Baltimore, Maryland
  - Beth Israel Deaconness Medical Center, Boston, Massachusetts
  - Advanced Rheumatology, Lansing, Michigan
  - Great Lakes Center of Rheumatology, Lansing, Michigan
  - Arthritis and Osteoporosis Associates of New Mexico, Las Cruces, New Mexico
  - Local Institution - 134, Great Neck, New York
  - North Shore-LIJ Health System-Division of Rheumatology, Great Neck, New York
  - NYU Langone Medical Center, New York, New York
  - Local Institution - 124, Syracuse, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - DJL Clinical Research, Charlotte, North Carolina
  - Local Institution - 101, Charlotte, North Carolina
  - Shanahan Rheumatology and Immunotherapy, Raleigh, North Carolina
  - MetroHealth Medical Systems, Cleveland, Ohio
  - St. Anthony's Medical Center, Oklahoma City, Oklahoma
  - Hershey Medical Center, Hershey, Pennsylvania
  - Local Institution - 136, Hershey, Pennsylvania
  - University of Pennsylvania Department of Dermatology, Philadelphia, Pennsylvania
  - University Of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh UPMC Lupus Center of Excellence, Pittsburgh, Pennsylvania
  - Advanced Rheumatology & Arthritis Research Center, PC, Wexford, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - Pioneer Research Solutions, Houston, Texas
  - Virginia Mason Medical Center, Seattle, Washington
- Argentina (14):
  - Local Institution - 628, Buenos Aires
  - Organización Médica de Investigación, Buenos Aires
  - Hospital General de Agudos Dr. Jose Maria Ramos Mejia, Buenos Aires
  - Local Institution - 625, Buenos Aires
  - Hospital Britanico de Buenos Aires, Buenos Aires
  - Consultora Integral de Salud Centro Médico Privado, Córdoba
  - Local Institution - 626, Córdoba
  - Hospital Privado Centro Medico de Cordoba, Córdoba
  - CER Instituto Mèdico, Quilmes
  - Local Institution - 630, Quilmes
  - Instituto de Investigaciones Clinicas de Quilmes, Quilmes
  - Local Institution - 629, Quilmes
  - Centro Medico Privado de Reumatologia, San Miguel de Tucumán
  - Local Institution - 627, San Miguel de Tucumán
- Belgium (6):
  - Hopital Erasme, Brussels
  - Local Institution - 425, Brussels
  - Local Institution - 427, Leuven
  - Universitaire Ziekenhuizen (UZ) Leuven - Gasthuisberg, Leuven
  - CHU de Liege, Liège
  - Local Institution - 426, Liège
- Brazil (13):
  - Centro Internacional de Pesquisas, Goiânia, Goiás
  - Local Institution - 655, Goiânia, Goiás
  - Centro de Estudos em Terapias Inovadoras LTDA, Curitiba, Paraná
  - Local Institution - 653, Curitiba, Paraná
  - LMK Servicos Medicos S/S, Porto Alegre, Rio Grande do Sul
  - Local Institution - 650, Porto Alegre, Rio Grande do Sul
  - Local Institution - 657, Campinas, São Paulo
  - State University of Campinas UNICAMP, Campinas, São Paulo
  - Local Institution - 652, Belo Horizonte
  - Santa Casa de Misericórdia de Belo Horizonte, Belo Horizonte
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, RS
  - Centro de Imunoterapia de Ipanema (CITIPA), Rio de Janeiro
  - Local Institution - 651, Rio de Janeiro
- Canada (12):
  - Local Institution - 205, Calgary, Alberta
  - The University of Calgary, Calgary, Alberta
  - Local Institution - 204, Winnipeg, Manitoba
  - University of Manitoba, Winnipeg, Manitoba
  - Local Institution - 201, Hamilton, Ontario
  - MAC Research Incorporated, Hamilton, Ontario
  - Local Institution - 202, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - CHUL du CHU de Quebec, Québec
  - Local Institution - 203, Québec
  - Clinique de Rhumatologie Du Centre Du Quebec, Québec
  - Local Institution - 200, Québec
- Colombia (15):
  - IPS Centro Integral de Reumatologia del Caribe Circaribe S.A.S., Barranquilla
  - Local Institution - 675, Barranquilla
  - Centro de Investigacion en Reumatologia y Especialidades Medicas S.A.S. - Cireem S.A.S, Bogotá
  - Local Institution - 682, Bogotá
  - Idearg S.A.S., Bogotá
  - Local Institution - 676, Bogotá
  - Local Institution - 679, Bucaramanga
  - Medicity S.A.S., Bucaramanga
  - Servimed S.A.S., Bucaramanga
  - Local Institution - 677, Chía
  - Preventive Care, Chía
  - Local Institution - 678, Medellín
  - Reumalab - Centro Integral de Reumatologia, Medellín
  - Hospital Pablo Tobon Uribe, Medellín
  - Local Institution - 680, Medellín
- France (4):
  - CHRU de Lille France, Lille
  - Assistance Publique - Hopitaux de Paris - Hopital Universitaire Pitie Salpetriere, Paris
  - Local Institution - 326, Paris
  - CHU Hautepierre, Strasbourg
- Germany (5):
  - Local Institution - 300, Cologne
  - Universitaetsklinikum Koeln, Cologne
  - Local Institution - 302, Kiel
  - Universitatsklinikum Schleswig-Holstein, Kiel
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
- Hungary (6):
  - Local Institution - 352, Budapest
  - Qualiclinic kft, Budapest
  - Egyesitett Szent Istvan es Szent Laszlo Korhaz - Rendelointezet, Budapest
  - Local Institution - 350, Budapest
  - Bekes Megyei Kozponti Korhaz, Gyula
  - Local Institution - 351, Gyula
- Italy (3):
  - ASST Spedali Civili P.O. di Brescia, Brescia
  - University of Ferrara, Azienda Ospedaliera-Universitaria S.Anna, Ferrara
  - Azienda Ospedaliero - Universitaria di Cagliari, Monserrato
- Mexico (16):
  - Centro de Investigacion en Artritis y Osteoporosis, Mexicali, Estado de Baja California
  - Local Institution - 610, Mexicali, Estado de Baja California
  - Centro Integral en Reumatología, S.A. de C.V., Guadalajara, Jalisco
  - Local Institution - 600, Guadalajara, Jalisco
  - Biológicos Especializados S.A. de C.V., Mexico City, Mexico City
  - Local Institution - 602, Mexico City, Mexico City
  - Clinica Integral de Osteoporosis y Artitis Reumatoide CLINOSAR, Mexico City, Mexico City
  - Local Institution - 608, Mexico City, Mexico City
  - Centro de Investigación y Tratamiento Reumatológico, Mexico City, Mexico City
  - Local Institution - 607, Mexico City, Mexico City
  - Centro de Alta Especialidad en Reumatología e Investigación del Potosí S.C., San Luis Potosí City, San Luis Potosí
  - Local Institution - 603, San Luis Potosí City, San Luis Potosí
  - Local Institution - 605, Mérida, Yucatán
  - Unidad de Atencion Medica e Investigacion en Salud, S.C., Mérida, Yucatán
  - Hospital Angeles Lindavista, D.F, DF
  - Local Institution - 606, D.F, DF
- Poland (10):
  - Local Institution - 380, Wroclaw, Woj. Dolnoslaskie
  - Local Institution - 377, Bydgoszcz
  - Szpital Uniwersytecki nr 2 im. Dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Local Institution - 376, Kościan
  - Samodzielny Publiczny Zespól Opieki Zdrowotnej w Koscianie Szpital im. Teodora Dunina, Kościan
  - Centrum Medyczne Plejady, Krakow
  - Local Institution - 375, Krakow
  - Local Institution - 378, Lublin
  - Samodzielny Publiczny Szpital Kliniczny nr 4, Klinika Reumatologii i Ukladowych Chorob Tkanki Laczne, Lublin
  - Niepubliczny Zaklad Opieki Zdrowotnej Biogenes Sp. z o.o., Wroclaw
- Russia (16):
  - City Clinical Hospital, Kazan'
  - Local Institution - 506, Kazan'
  - Kemerovo State Medical Academy, Kemerovo
  - Local Institution - 505, Kemerovo
  - Institution of the Russian Academy of Medical Sciences Research Institute of Rheumatology of the Ru, Moscow
  - Local Institution - 507, Moscow
  - Local Institution - 500, Orenburg
  - Orenburg State Medical Academy, Orenburg
  - Saint Petersburg Research Institute for Emergency Medical Care, Saint Petersburg
  - Leningrad Regional Clinical Hospital, Saint Petersburg
  - Local Institution - 502, Saint Petersburg
  - Local Institution - 503, Saint Petersburg
  - State Higher Educational Institution, Saint Petersburg
  - BioMed, LLC., Vladimir
  - Local Institution - 504, Vladimir
  - Voronezh Regional Clinical Hopsital #1, Voronezh State Medical Academy, Voronezh
- Serbia (10):
  - Institute of Rheumatology Belgrade, Belgrade
  - Local Institution - 475, Belgrade
  - Local Institution - 476, Belgrade
  - Local Institution - 477, Belgrade
  - Local Institution - 478, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - Local Institution - 480, Kragujevac
  - Institute Niska Banja, Niška Banja
  - Local Institution - 479, Niška Banja
- Spain (8):
  - Hospital Universitario a Coruna, A Coruña
  - Local Institution - 400, A Coruña
  - Hospital Universitario Vall D hebron, Barcelona
  - Local Institution - 403, Barcelona
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital Marques de Valdecilla, Santander
  - Local Institution - 405, Santander
  - Hospital Universitario Araba - Txagorritxu, Vitoria-Gasteiz

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nakayama Y, Kosek J, Capone L, Hur EM, Schafer PH, Ringheim GE. Aiolos Overexpression in Systemic Lupus Erythematosus B Cell Subtypes and BAFF-Induced Memory B Cell Differentiation Are Reduced by CC-220 Modulation of Cereblon Activity. J Immunol. 2017 Oct 1;199(7):2388-2407. doi: 10.4049/jimmunol.1601725. Epub 2017 Aug 28. PMID 28848067
- [Derived] Lipsky PE, Vollenhoven RV, Dorner T, Werth VP, Merrill JT, Furie R, Petronijevic M, Velasco Zamora B, Majdan M, Irazoque-Palazuelos F, Terbrueggen R, Delev N, Weiswasser M, Korish S, Stern M, Hersey S, Ye Y, Gaudy A, Liu Z, Gagnon R, Tang S, Schafer PH. Biological impact of iberdomide in patients with active systemic lupus erythematosus. Ann Rheum Dis. 2022 Jul 12;81(8):1136-1142. doi: 10.1136/annrheumdis-2022-222212. PMID 35477518
- [Derived] Merrill JT, Werth VP, Furie R, van Vollenhoven R, Dorner T, Petronijevic M, Velasco J, Majdan M, Irazoque-Palazuelos F, Weiswasser M, Korish S, Ye Y, Gaudy A, Schafer PH, Liu Z, Agafonova N, Delev N. Phase 2 Trial of Iberdomide in Systemic Lupus Erythematosus. N Engl J Med. 2022 Mar 17;386(11):1034-1045. doi: 10.1056/NEJMoa2106535. PMID 35294813
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- PBO QD: Placebo-matching treatment once a day.
- 0.45 mg QD: Participants dosed with CC-220 at 0.45 mg once a day
- 0.15 mg QD: Participants dosed with CC-220 at 0.15 mg once a day
- 0.30 mg QD: Participants dosed with CC-220 at 0.30 mg once a day
Period: Placebo Controlled Phase
Arm/Group | PBO QD | 0.45 mg QD | 0.15 mg QD | 0.30 mg QD
Started | 83 | 82 | 42 | 82
Completed | 83 | 81 | 42 | 82
Not Completed | 0 | 1 | 0 | 0
Not completed — Participant Withdrew Consent | 0 | 1 | 0 | 0
Period: Treatment Period
Arm/Group | PBO QD | 0.45 mg QD | 0.15 mg QD | 0.30 mg QD
Started (Started = Entered placebo-controlled phase) | 83 | 81 | 42 | 82
Going to 0.30mg After Week 24 (After Week 24) | 36 | 0 | 0 | 0
Going to 0.45mg After Week 24 | 36 | 0 | 0 | 0
Staying on Placebo After Week 24 | 11 | 0 | 0 | 0
Completed (Completed = Finished placebo-controlled phase) | 73 | 73 | 39 | 62
Not Completed | 10 | 8 | 3 | 20
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 2 | 1 | 11
Not completed — Pregnancy | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 5 | 2 | 6
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Other reasons | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PBO QD | 0.15 mg QD | 0.30 mg QD | 0.45 mg QD | Total
Number analyzed (Participants) | 83 | 42 | 82 | 82 | 289
Age, Customized [Count of Participants; unit: Participants]
  < 40 years old | 33 | 15 | 31 | 25 | 104
  >= 40 to <= 50 | 26 | 15 | 21 | 28 | 90
  > 50 to < 65 | 19 | 10 | 24 | 24 | 77
  >= 65 | 5 | 2 | 6 | 5 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 41 | 77 | 80 | 279
  Male | 2 | 1 | 5 | 2 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 21 | 46 | 33 | 141
  Not Hispanic or Latino | 42 | 21 | 36 | 49 | 148
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 5 | 1 | 5 | 13
  Asian | 0 | 0 | 1 | 0 | 1
  Black or African American | 7 | 3 | 6 | 5 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  White | 60 | 29 | 59 | 61 | 209
  Not collected or reported | 0 | 0 | 0 | 0 | 0
  Other | 14 | 5 | 15 | 11 | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieve SLE Responder Index (SRI) (4) Response
Description: The primary objective is to evaluate the clinical efficacy of three doses of CC-220 (0.45 mg once per day [QD], 0.3 mg QD or 0.15 mg QD) compared to placebo, for the treatment of active systemic lupus erythematosus (SLE) using the SLE Responder Index at Week 24 Composite endpoint SRI(4), defined by the following criteria: - Reduction from Baseline of ≥ 4 points in the Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) 2K score and - No new one or more British Isles Lupus Assessment Group (BILAG) A or new (excludes A to B) 2 or more BILAG B items compared to Baseline using BILAG 2004 Index and - No worsening from Baseline defined by an increase of < 0.30 points from Baseline on a Physician's Global Assessment (PGA) visual analog scale (VAS) from 0-3
Time Frame: Week 24
Population: Primary analysis based on Intent-to-treat (ITT) Population (all randomized participants who received at least one dose of investigational product) and nonresponder imputation (NRI). Participants with insufficient data for response determination at the given time point are considered nonresponders.
Measure: Number; unit: Number of participants
Arm/Group | PBO QD | 0.15 mg QD | 0.30 mg QD | 0.45 mg QD
Number analyzed (Participants) | 83 | 42 | 82 | 81
Number of participants | 29 | 20 | 33 | 44
Statistical Analysis 1: Comparison: PBO QD vs 0.15 mg QD; Test type: Superiority; p = 0.214, Cochran-Mantel-Haenszel; Stratified difference = 11.4, 95% CI 2-sided [-6.57 to 29.00]
Statistical Analysis 2: Comparison: PBO QD vs 0.30 mg QD; Test type: Superiority; p = 0.512, Cochran-Mantel-Haenszel; Stratified difference = 5.0, 95% CI 2-sided [-9.77 to 19.48]
Statistical Analysis 3: Comparison: PBO QD vs 0.45 mg QD; Test type: Superiority; p = 0.011, Cochran-Mantel-Haenszel; Stratified difference = 19.4, 95% CI 2-sided [4.12 to 33.42]

2. Secondary Outcome: Number of Participants With SLEDAI 2K Score Improvement of ≥ 4 Points From Baseline
Description: The SLEDAI 2K score measures disease activity through assessment of 24 lupus manifestations using a weighted score of 1 to 8 points. A manifestation is recorded if it is present over the previous 30 days regardless of severity or whether it has improved or worsened. A SLEDAI 2K score of 3 to 4 points is representative of active disease and a decrease of 1 to 2 points is considered clinically meaningful.
Time Frame: Week 24
Population: ITT population. Participants with insufficient data for response determination at the given time point are considered nonresponders.
Measure: Number; unit: Number of participants
Arm/Group | PBO QD | 0.15 mg QD | 0.30 mg QD | 0.45 mg QD
Number analyzed (Participants) | 83 | 42 | 82 | 81
Number of participants | 30 | 20 | 35 | 45
Statistical Analysis 1: Comparison: PBO QD vs 0.15 mg QD; Test type: Superiority; p = 0.264, Cochran-Mantel-Haenszel; Stratified difference = 10.3, 95% CI 2-sided [-7.66 to 27.97]
Statistical Analysis 2: Comparison: PBO QD vs 0.30 mg QD; Test type: Superiority; p = 0.399, Cochran-Mantel-Haenszel; Stratified difference = 6.5, 95% CI 2-sided [-8.45 to 21.00]
Statistical Analysis 3: Comparison: PBO QD vs 0.45 mg QD; Test type: Superiority; p = 0.012, Cochran-Mantel-Haenszel; Stratified difference = 19.3, 95% CI 2-sided [4.01 to 33.36]

3. Secondary Outcome: Number of Participants With a ≥ 50% Reduction in Cutaneous Lupus Area and Severity Index (CLASI) Activity Score From Baseline, in Participants With Baseline CLASI Activity Score ≥ 10
Description: The CLASI Activity Score ranges from 0 to 70. To generate the activity score erythema is scored on a scale of 0 (absent) to 3 (dark red; purple/violaceous/crusted/hemorrhagic) and scale/hypertrophy are scored on a scale of 0 (absent) to 2 (verrucous/hypertrophic). Both the erythema and scale/hypertrophy scores are assessed in 13 different anatomical locations. In addition, the presence of mucous membrane lesions is scored on a scale of 0 (absent) to 1 (lesion or ulceration), the occurrence of recent hair loss is captured (1=yes; 0=no) and non-scarring alopecia is scored on a scale of 0 (absent) to 3 (focal or patchy in more than one quadrant). To calculate the activity score, all scores for erythema, scale/hypertrophy, mucous membrane lesions and alopecia are added together.
Time Frame: Week 24
Population: ITT population with Baseline CLASI activity score ≥ 10
Measure: Number; unit: Number of participants
Arm/Group | PBO QD | 0.15 mg QD | 0.30 mg QD | 0.45 mg QD
Number analyzed (Participants) | 16 | 11 | 18 | 19
Number of participants | 8 | 8 | 8 | 13
Statistical Analysis 1: Comparison: PBO QD vs 0.15 mg QD; Test type: Superiority; p = 0.446, Cochran-Mantel-Haenszel; Stratified difference = 24.0, 95% CI 2-sided [-12.38 to 53.11]
Statistical Analysis 2: Comparison: PBO QD vs 0.30 mg QD; Test type: Superiority; p > 0.999, Cochran-Mantel-Haenszel; Stratified difference = 5.3, 95% CI 2-sided [-27.64 to 39.38]
Statistical Analysis 3: Comparison: PBO QD vs 0.45 mg QD; Test type: Superiority; p = 0.488, Cochran-Mantel-Haenszel; Stratified difference = 14.2, 95% CI 2-sided [-19.54 to 44.48]

4. Secondary Outcome: Number of Participants With no New Organ System Affected as Defined by 1 or More BILAG A or New (Excludes A to B) 2 or More BILAG B Items Compared to Baseline Using BILAG 2004 Index
Description: The BILAG 2004 is a composite index that is based on the Classic BILAG index. It is a clinical measure of lupus disease activity. This tool assesses the changing severity of clinical manifestations of SLE using an ordinal scale scoring system that contain 9 systems (constitutional, mucocutaneous, neuropsychiatric, musculoskeletal, cardiorespiratory, gastrointestinal, ophthalmic, renal and hematological). Activity in each organ system is scored as: A=most active disease; B=intermediate activity; C=mild, stable disease; D=previous involvement, currently inactive; E=no previous activity.
Time Frame: Week 24
Population: All treated participants
Measure: Number; unit: Number of participants
Arm/Group | PBO QD | 0.15 mg QD | 0.30 mg QD | 0.45 mg QD
Number analyzed (Participants) | 83 | 42 | 82 | 81
Number of participants | 65 | 38 | 59 | 70
Statistical Analysis 1: Comparison: PBO QD vs 0.15 mg QD; Test type: Superiority; p = 0.092, Cochran-Mantel-Haenszel; Stratified difference = 12.4, 95% CI 2-sided [-2.74 to 24.07]
Statistical Analysis 2: Comparison: PBO QD vs 0.30 mg QD; Test type: Superiority; p = 0.434, Cochran-Mantel-Haenszel; Stratified difference = -5.3, 95% CI 2-sided [-18.43 to 8.06]
Statistical Analysis 3: Comparison: PBO QD vs 0.45 mg QD; Test type: Superiority; p = 0.182, Cochran-Mantel-Haenszel; Stratified difference = 8.0, 95% CI 2-sided [-3.88 to 19.65]

5. Secondary Outcome: Percentage of Participants With no Worsening (Increase of < 0.30 Points From Baseline) in PGA Compared to Baseline
Description: The PGA uses a visual analog scale with scores between 0 and 3 to indicate worsening of disease. The scoring is as follows: 0 = none, 1 = mild disease, 2 = moderate disease, and 3 = severe disease.
Time Frame: Week 24
Population: All treated participants
Measure: Number; unit: Percentage of participants
Arm/Group | PBO QD | 0.15 mg QD | 0.30 mg QD | 0.45 mg QD
Number analyzed (Participants) | 83 | 42 | 82 | 81
Percentage of participants | 78.3 | 90.5 | 73.2 | 85.2
Statistical Analysis 1: Comparison: PBO QD vs 0.15 mg QD; Test type: Superiority; p = 0.098, Cochran-Mantel-Haenszel; Stratified difference = 12.1, 95% CI 2-sided [-2.98 to 23.78]
Statistical Analysis 2: Comparison: PBO QD vs 0.30 mg QD; Test type: Superiority; p = 0.521, Cochran-Mantel-Haenszel; Stratified difference = -4.3, 95% CI 2-sided [-17.36 to 8.92]
Statistical Analysis 3: Comparison: PBO QD vs 0.45 mg QD; Test type: Superiority; p = 0.267, Cochran-Mantel-Haenszel; Stratified difference = 6.8, 95% CI 2-sided [-5.24 to 18.55]

6. Secondary Outcome: Mean Change From Baseline in Swollen Joint Count in Participants With ≥ 2 Swollen Joints at Baseline
Description: Joint tenderness and swelling will be noted as "present" or "absent," with no quantitation of severity using a 28- joint count. Note: Data presented is Adjusted mean data.
Time Frame: Week 24
Population: ITT Population; Subjects with >=2 Swollen Joints, with a baseline value and a value at the time point.
Measure: Mean (95% Confidence Interval); unit: swollen joints
Arm/Group | PBO QD | 0.15 mg QD | 0.30 mg QD | 0.45 mg QD
Number analyzed (Participants) | 62 | 33 | 54 | 56
swollen joints | -6.7 [-7.2 to -6.2] | -6.0 [-6.7 to -5.3] | -6.0 [-6.7 to -5.2] | -6.6 [-7.1 to -6.1]
Statistical Analysis 1: Comparison: PBO QD vs 0.15 mg QD; Test type: Superiority; p = 0.116, longitudinal data analysis model; Difference in adjusted mean = 0.7, 95% CI 2-sided [-0.2 to 1.5]
Statistical Analysis 2: Comparison: PBO QD vs 0.30 mg QD; Test type: Superiority; p = 0.094, longitudinal data analysis model; Difference in adjusted mean = 0.7, 95% CI 2-sided [-0.1 to 1.6]
Statistical Analysis 3: Comparison: PBO QD vs 0.45 mg QD; Test type: Superiority; p = 0.881, longitudinal data analysis model; Difference in adjusted mean = 0.1, 95% CI 2-sided [-0.6 to 0.8]

7. Secondary Outcome: Mean Change From Baseline in Tender Joint Count in Participants With ≥ 2 Tender Joints at Baseline
Description: as for outcome 6
Time Frame: Week 24
Population: ITT Population; Participants with >=2 Tender Joints, with a baseline value and a value at the time point.
Measure: Mean (95% Confidence Interval); unit: tender joints
Arm/Group | PBO QD | 0.15 mg QD | 0.30 mg QD | 0.45 mg QD
Number analyzed (Participants) | 62 | 33 | 54 | 56
tender joints | -7.9 [-8.8 to -7.0] | -6.8 [-8.1 to -5.6] | -6.7 [-7.7 to -5.6] | -7.6 [-8.5 to -6.7]
Statistical Analysis 1: Comparison: PBO QD vs 0.15 mg QD; Test type: Superiority; p = 0.160, longitudinal data analysis model; Difference in adjusted mean = 1.1, 95% CI 2-sided [-0.4 to 2.6]
Statistical Analysis 2: Comparison: PBO QD vs 0.30 mg QD; Test type: Superiority; p = 0.056, longitudinal data analysis model; Difference in adjusted mean = 1.3, 95% CI 2-sided [0.0 to 2.6]
Statistical Analysis 3: Comparison: PBO QD vs 0.45 mg QD; Test type: Superiority; p = 0.621, longitudinal data analysis model; Difference in adjusted mean = 0.3, 95% CI 2-sided [-1.0 to 1.6]

8. Secondary Outcome: Mean Change From Baseline in PGA Score
Description: as for outcome 5
Time Frame: Week 24
Population: ITT population with a baseline value and a value at the time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | PBO QD | 0.15 mg QD | 0.30 mg QD | 0.45 mg QD
Number analyzed (Participants) | 66 | 38 | 63 | 70
scores on a scale | -0.803 (0.605) | -0.805 (0.528) | -0.819 (0.629) | -0.883 (0.546)

9. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Score
Description: The FACIT-Fatigue scale is a 13-item self-administered questionnaire that assesses both the physical and functional consequences of fatigue. Each question is answered on a 5-point scale, where 0 means "not at all," and 4 means "very much." The total FACIT-Fatigue score ranges from 0 to 52. Note: Data presented is Adjusted mean data.
Time Frame: Week 24
Population: ITT population; participants with a baseline value and a value at the time point
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | PBO QD | 0.15 mg QD | 0.30 mg QD | 0.45 mg QD
Number analyzed (Participants) | 67 | 38 | 60 | 69
scores on a scale | 3.8 [1.6 to 6.0] | 2.7 [-0.3 to 5.6] | 3.1 [0.9 to 5.4] | 5.2 [3.0 to 7.4]
Statistical Analysis 1: Comparison: PBO QD vs 0.15 mg QD; Test type: Superiority; p = 0.546, longitudinal data analysis model; Difference in adjusted mean = -1.1, 95% CI 2-sided [-4.7 to 2.5]
Statistical Analysis 2: Comparison: PBO QD vs 0.30 mg QD; Test type: Superiority; p = 0.681, longitudinal data analysis model; Difference in adjusted mean = -0.6, 95% CI 2-sided [-3.7 to 2.4]
Statistical Analysis 3: Comparison: PBO QD vs 0.45 mg QD; Test type: Superiority; p = 0.350, longitudinal data analysis model; Difference in adjusted mean = 1.4, 95% CI 2-sided [-1.6 to 4.4]

10. Secondary Outcome: Percentage of Participants With Corticosteroid Reduction
Description: - The percentage of participants with a prednisone or equivalent dose of ≥ 10 mg/day at Baseline whose prednisone or equivalent dose has been reduced to ≤ 7.5 mg/day by Week 16 and maintained through Week 24 with no flares between Week 16 and Week 24 - The percentage of participants with a prednisone or equivalent dose of ≥ 10 mg/day at Baseline whose prednisone or equivalent dose has been reduced to < 10 mg/day by Week 16 and maintained through Week 24 with no flares between Week 16 and Week 24
Time Frame: Week 24
Population: ITT Population; Participants with Baseline OCS Dose >= 10 mg/day Participants with insufficient data for response determination at the given time point are considered nonresponders.
Measure: Number; unit: Percentage of participants
Arm/Group | PBO QD | 0.15 mg QD | 0.30 mg QD | 0.45 mg QD
Number analyzed (Participants) | 31 | 17 | 30 | 32
Percentage of participants
  Week 24, <= 7.5 mg/day | 3.2 | 0.0 | 3.3 | 0.0
  Week 24, < 10 mg/day | 6.5 | 0.0 | 3.3 | 0.0
Statistical Analysis 1: Comparison: PBO QD vs 0.30 mg QD; Test type: Superiority — <= 7.5 mg/day; p > 0.999, longitudinal data analysis model; Stratified difference = 0.2, 95% CI 2-sided [-15.13 to 15.91]
Statistical Analysis 2: Comparison: PBO QD vs 0.30 mg QD; Test type: Superiority — < 10 mg/day; p > 0.999, longitudinal data analysis model; Stratified difference = -3.2, 95% CI 2-sided [-17.74 to 13.00]

11. Secondary Outcome: Percent Change From Baseline in Corticosteroid Reduction
Description: Percent change from Baseline in oral corticosteroid (OCS) dose in subjects with prednisone or equivalent ≥ 10 mg/day at Baseline Note: Data presented is Adjusted mean data.
Time Frame: Week 24
Population: ITT Population; Participants with the Baseline OCS Dose >= 10 mg/day, with a baseline value and a value at the time point.
Measure: Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | PBO QD | 0.15 mg QD | 0.30 mg QD | 0.45 mg QD
Number analyzed (Participants) | 26 | 17 | 25 | 30
percent change from baseline | -7.9 [-13.6 to -2.2] | -5.1 [-11.9 to 1.6] | -3.8 [-9.5 to 2.0] | -1.4 [-6.4 to 3.6]
Statistical Analysis 1: Comparison: PBO QD vs 0.15 mg QD; Test type: Superiority; p = 0.535, longitudinal data analysis model; Difference in adjusted means = 2.8, 95% CI 2-sided [-6.0 to 11.6]
Statistical Analysis 2: Comparison: PBO QD vs 0.30 mg QD; Test type: Superiority; p = 0.309, longitudinal data analysis model; Difference in adjusted means = 4.2, 95% CI 2-sided [-3.9 to 12.2]
Statistical Analysis 3: Comparison: PBO QD vs 0.45 mg QD; Test type: Superiority; p = 0.091, longitudinal data analysis model; Difference in adjusted means = 6.5, 95% CI 2-sided [-1.0 to 14.1]

12. Secondary Outcome: The Total Corticosteroid Dose From Baseline Through Week 24
Description: Standardized total oral corticosteroid (OCS) dose.
Time Frame: Through Week 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | PBO QD | 0.15 mg QD | 0.30 mg QD | 0.45 mg QD
Number analyzed (Participants) | 83 | 42 | 82 | 81
mg | 1139.7 (916.9) | 1101.9 (827.1) | 1071.8 (965.0) | 1105.5 (969.3)

13. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Number of participants who experienced a TEAE during the course of the study
Time Frame: from first dose to 28 days post-last dose through Week 24 (placebo-controlled phase), approximately 28 weeks total
Population: All treated participants
Measure: Number; unit: Number of participants
Arm/Group | PBO QD | 0.15 mg QD | 0.30 mg QD | 0.45 mg QD
Number analyzed (Participants) | 83 | 42 | 82 | 81
Number of participants
  Any TEAE | 54 | 31 | 64 | 63
  Any Drug-related TEAE | 24 | 14 | 36 | 32
  Any Serious TEAE | 7 | 3 | 4 | 6
  Any Severe TEAE | 5 | 3 | 4 | 1
  Any TEAE Leading to Drug Interruption | 15 | 10 | 14 | 23
  Any TEAE Leading to Drug Withdrawal | 6 | 2 | 11 | 4
  Any TEAE Leading to Death | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: The number at Risk for All-Cause Mortality represents all Randomized Participants; From date of randomization to 100 days post last dose. Approximately Up to 47 Months The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication; 28 days post last dose Approximately up to 48 months
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Groups:
- 0.15mg QD: Participants dosed with CC-220 at 0.15 mg once a day
- 0.30mg QD; Active Treatment Phase 0.30mg Following Placebo: Participants dosed with CC-220 at 0.30 mg once a day
- 0.45mg QD; Active Treatment Phase 0.45mg Following Placebo: Participants dosed with CC-220 at 0.45 mg once a day
- Placebo: Placebo-matching treatment once a day.
Arm/Group | 0.15mg QD | 0.30mg QD | 0.45mg QD | Placebo | Active Treatment Phase 0.30mg Following Placebo | Active Treatment Phase 0.45mg Following Placebo
All-Cause Mortality (participants affected / at risk) | 1/42 | 0/82 | 0/81 | 1/83 | 1/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 6/42 | 10/82 | 14/81 | 7/83 | 2/36 | 3/36
Other Adverse Events (participants affected / at risk) | 32/42 | 63/82 | 62/81 | 34/83 | 16/36 | 26/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.15mg QD (N=42) | 0.30mg QD (N=82) | 0.45mg QD (N=81) | Placebo (N=83) | Active Treatment Phase 0.30mg Following Placebo (N=36) | Active Treatment Phase 0.45mg Following Placebo (N=36)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Implant site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 3 | 0 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Varicella zoster pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Suture related complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Joint instability (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 0 | 0
Brain stem infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abnormal uterine bleeding (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 3 | 0 | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.15mg QD (N=42) | 0.30mg QD (N=82) | 0.45mg QD (N=81) | Placebo (N=83) | Active Treatment Phase 0.30mg Following Placebo (N=36) | Active Treatment Phase 0.45mg Following Placebo (N=36)
Anaemia (Blood and lymphatic system disorders) | 3 | 5 | 6 | 2 | 3 | 2
Leukopenia (Blood and lymphatic system disorders) | 3 | 3 | 10 | 1 | 4 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 4 | 1 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 8 | 16 | 2 | 2 | 4
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2 | 1 | 3 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 6 | 5 | 8 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 3 | 4 | 5 | 2 | 0 | 1
Vomiting (Gastrointestinal disorders) | 6 | 5 | 3 | 2 | 1 | 1
Pyrexia (General disorders) | 3 | 1 | 3 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 4 | 6 | 5 | 3 | 1 | 1
COVID-19 (Infections and infestations) | 0 | 2 | 3 | 0 | 2 | 1
Gastroenteritis (Infections and infestations) | 0 | 3 | 3 | 1 | 2 | 0
Influenza (Infections and infestations) | 4 | 5 | 8 | 3 | 2 | 3
Nasopharyngitis (Infections and infestations) | 5 | 7 | 10 | 1 | 4 | 3
Oral herpes (Infections and infestations) | 4 | 1 | 2 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 5 | 6 | 4 | 1 | 1 | 1
Sinusitis (Infections and infestations) | 1 | 5 | 5 | 1 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 6 | 11 | 15 | 4 | 3 | 6
Urinary tract infection (Infections and infestations) | 7 | 24 | 15 | 3 | 2 | 6
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 0 | 1 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 3 | 2 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 5 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 3 | 1
Dizziness (Nervous system disorders) | 0 | 4 | 0 | 2 | 1 | 3
Headache (Nervous system disorders) | 3 | 3 | 4 | 5 | 2 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 1 | 2 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 4 | 0 | 2 | 0
Hypertension (Vascular disorders) | 2 | 4 | 5 | 2 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT03161483/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/83/NCT03161483/SAP_001.pdf